CLINICAL TRIAL: NCT00980941
Title: The Effect of Different Types of Starch on Glycemic Response, Subjective Appetite and Short-term Food Intake in Young Men
Brief Title: Types of Starch and Their Effect on Blood Glucose, Appetite and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Ingredion Incorporated (Industry)
Responsible Party: G. Harvey Anderon, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Starch study 1; National Starch_ethics_21513
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Obesity Prevention; Diabetes Prevention
Keywords: starch; carbohydrates; blood glucose; food intake; satiety; appetite
MeSH Terms: interventions — Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Soup with no added starch (Experimental)
  Interventions: Dietary Supplement: soup with or without starch
- Soup + 50 g of whole grain starch (Experimental)
  Interventions: Dietary Supplement: soup with or without starch
- Soup + 50 g of high amylose corn starch (Experimental)
  Interventions: Dietary Supplement: soup with or without starch
- Soup + 50 g of regular corn starch (Experimental)
  Interventions: Dietary Supplement: soup with or without starch
- Soup + 50 g maltodextrin starch (Experimental)
  Interventions: Dietary Supplement: soup with or without starch

INTERVENTIONS:
Dietary Supplement: soup with or without starch

SUMMARY:
The investigators hypothesize that different types of starch vary in their effects on appetite, blood sugar and food intake. In this study, subjects consumed five soups containing 50 g of whole grain, high amylose corn, regular corn or maltodextrin starches or no added starch at one week intervals. The investigators measured food intake at 30 minutes, appetite and blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males with a BMI of 20-24.9 kg/m2

Exclusion Criteria:

* Females
* Smokers
* Breakfast skippers
* Individuals with diabetes or other metabolic diseases

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 0-170 min
Food intake | at 30 min after the treatment
Appetite | 0-170 min

SECONDARY OUTCOMES:
Water intake | at 30 min
Palatability of treatments | 0-170 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Studies, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Anderson GH, Cho CE, Akhavan T, Mollard RC, Luhovyy BL, Finocchiaro ET. Relation between estimates of cornstarch digestibility by the Englyst in vitro method and glycemic response, subjective appetite, and short-term food intake in young men. Am J Clin Nutr. 2010 Apr;91(4):932-9. doi: 10.3945/ajcn.2009.28443. Epub 2010 Feb 17. PMID 20164321